CLINICAL TRIAL: NCT07385924
Title: Evaluation of Accuracy of the Use of 3d Printed Reduction Guide in Treatment of Mandibular Fractures Using Two Different Methods of Virtual Planning
Brief Title: Evaluation of the Accuracy of 3d Printed Reduction Guide in Treatment of Mandibular Fractures Using Two Different Methods of Virtual Planning
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00010825-12/2023
Record Dates: First submitted 2026-01-19; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Mandibular Fracture; Virtual Plan of Mandibular Fracture
Keywords: mandibular fracture; virtual surgical planning
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients were allocated in a 1:1 ratio using an on-site computer software system with concealed allocation through sequentially numbered, opaque, sealed envelopes (SNOSE). (group A) virtual planning will be done using the manual virtual reduction method and (group B) virtual planning will be done using the mirror image technique.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual planning will be done using the manual virtual reduction method (Experimental): virtual planning will be done using the manual virtual reduction method and . Design of the reduction guide will be done in accordance with the virtual plan. The surgical reduction will be done with the aid of the guide.
  Interventions: Device: Mandibular fracture treatment by 3d printed guide where virtual planning will be done using the manual reduction technique.
- virtual planning will be done using the mirror image technique. (Experimental): virtual planning will be done using the mirror image technique. Design of the reduction guide will be done in accordance with the virtual plan. The surgical reduction will be done with the aid of the guide.
  Interventions: Device: Mandibular fracture treatment by 3d printed guide where virtual planning will be done using the mirror image reduction technique.

INTERVENTIONS:
Device: Mandibular fracture treatment by 3d printed guide where virtual planning will be done using the manual reduction technique. — Mandibular fracture treatment by 3d printed guide where virtual planning will be done using the manual reduction technique.
  Arms: virtual planning will be done using the manual virtual reduction method
Device: Mandibular fracture treatment by 3d printed guide where virtual planning will be done using the mirror image reduction technique. — Mandibular fracture treatment by 3d printed guide where virtual planning will be done using the mirror image reduction technique.
  Arms: virtual planning will be done using the mirror image technique.

SUMMARY:
This study will evaluate the accuracy of the use of 3-D printed reduction guide in treatment of mandibular fractures using two different methods of virtual planning.

DETAILED DESCRIPTION:
This study will be conducted clinically on 24 patients with mandibular fracture divided into 2 groups, (group A) virtual planning will be done using the manual virtual reduction method and (group B) virtual planning will be done using the mirror image technique. Design of the reduction guide will be done in accordance with the virtual plan. The surgical reduction will be done with the aid of the guide.

ELIGIBILITY:
Inclusion Criteria:

* Medically fit patients free from relevant conditions contraindicating surgery.
* Unilateral mandibular fractures indicated for open reduction and internal fixation

Exclusion Criteria:

* Infected fracture site.
* Patients with systemic bone diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of accuracy of mandibular reduction of each surgical guide. | Immediately after the surgery
  Evaluation of accuracy of surgical guide will be done using slicer and blender software with the aid of the preoperative and postoperative CT.
  Preoperative planning will be merged with the new CT data to identify the accuracy of reduction.
  Landmark-Based Positional Analysis was used to quantify positional accuracy of the reduced mandibular segment. Bilateral mandibular landmarks were selected to represent the spatial position of the fractured and adjacent segments. The selected landmarks included condylion (Co), gonion (Go), and mental foramen (MF), which are distributed across the mandibular ramus, angle, and body regions. linear distances to the three reference planes were recorded in millimeters. To provide a comprehensive three-dimensional representation of positional discrepancy, an asymmetry index (AI) was calculated for each bilateral landmark.

SECONDARY OUTCOMES:
Clinical evaluation of postoperative occlusion | 3 months
  Assessment of occlusion will be done By checking the maximal intercuspal position (centric occlusion) to ensure proper occlusal relationship including molar relation, canine relation and midline centralization.
  The percentage of patients suffering from occlusal disturbances will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes